CLINICAL TRIAL: NCT06637631
Title: A Phase 2, Multinational, Multicenter, Randomized, Doubleblind, Placebocontrolled, Dose-ranging Study to Evaluate the Efficacy and Safety of SAR441566 in Adults With Moderate to Severe Crohn's Disease.
Brief Title: A Study to Investigate Efficacy and Safety of SAR441566 in Patients With Crohn's Disease.
Acronym: SPECIFI-CD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI18212; 2024-512633-32-00 (Registry Identifier: CTIS); U1111-1301-3830 (Other: WHO ICTRP)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAR441566 dose 1 (Experimental): Participants will receive SAR441566 dose 1.
  Interventions: Drug: SAR441566
- SAR441566 dose 2 (Experimental): Participants will receive SAR441566 dose 2.
  Interventions: Drug: SAR441566
- SAR441566 dose 3 (Experimental): Participants will receive SAR441566 dose 3.
  Interventions: Drug: SAR441566
- Placebo (Placebo Comparator): Participants will receive SAR441566 matching placebo.
  Interventions: Drug: SAR441566 matching Placebo

INTERVENTIONS:
Drug: SAR441566 — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: SAR441566 dose 1; SAR441566 dose 2; SAR441566 dose 3
Drug: SAR441566 matching Placebo — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: Placebo

SUMMARY:
This is a phase 2, multinational, multicenter, randomized, double-blind, placebo-controlled, dose-ranging study to evaluate the efficacy and safety of SAR441566 in adults with moderate to severe Crohn's Disease (CD). The primary objective of this study is to assess the efficacy of different doses of SAR441566 compared with placebo in participants with moderate to severe CD.

This study will have an anticipated duration of up to 59 weeks which will include a screening period of 4 weeks (+7 calendar days if needed), followed by the Main Study (MS) treatment period, lasting 52 weeks, and a 2-week follow-up period after end of treatment. The MS period includes a Double-Blind (DB) treatment period with 12 weeks of induction followed by 40 weeks of maintenance.

Additionally, an Open Label (OL) period of up to 40 weeks will be offered to eligible participants. The combined duration of the DB maintenance and OL periods cannot exceed 40 weeks, depending on when participants switch.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Male or female participants aged 18 to 75 years at the time of signing the ICF
2. Confirmed diagnosis of CD for at least 3 months prior to Baseline
3. Confirmed diagnosis of moderate to severe CD as assessed by:

   * Crohn's Disease Activity Index (CDAI) score and the Simple Endoscopic Score for Crohn's disease (SES-CD) on an endoscopy confirmed by a central reader
   * stool frequency (SF), abdominal pain (AP) score
4. History of prior exposure to standard treatment (5-ASA, steroids, immunomodulators or antibiotics) or advanced therapies (biologics or small molecules), but having inadequate response to, loss or response to or intolerance to at least one of these therapies
5. On stable doses of standard treatments prior to screening (Oral 5-ASA compounds, Oral corticosteroids, AZA, 6-MP, or MTX ..)
6. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Women participants should not be pregnant or breastfeeding.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Participants with active UC, indeterminate colitis or short bowel syndrome
2. Participants with CD isolated to the stomach, duodenum, jejunum, or peri anal region, without colonic or ileal involvement
3. Participants with following ongoing known complications of CD: fistula, abscess, symptomatic stricture/stenosis, fulminant colitis, toxic megacolon, recent bowel resection within 3 months of screening or history of > 3 bowel resections
4. Participants with stool sample positive for infectious pathogens
5. Participants with active tuberculosis (TB) or a history of incompletely treated active or latent TB per local guidelines
6. Participants with Positive Hepatitis B surface antigen (HBsAg) or positive Hepatitis B core antibody (HBcAb); and/or positive Hepatitis C antibody (HCV) at the Screening Visit
7. Participants with any other active, chronic or recurrent infection, including recurrent or disseminated herpes zoster or disseminated herpes simplex
8. Participants with a known history of Human Immunodeficiency Virus (HIV) infection or positive HIV-1 or HIV-2 serology at screening
9. Participants presenting with active malignancies, lymphoproliferative disease, or recurrence of either, within the 5 years before screening
10. History of colonic mucosal dysplasia or presence of colonic mucosal dysplasia or adenomatous colonic polyps not removed during colonoscopy at screening visit
11. Infection(s) requiring treatment with IV anti infectives within 30 days or oral/intramuscular anti-infectives within 14 days prior to the screening visit
12. Participants requiring or receiving any parental nutrition and/or exclusive enteral nutrition
13. Participants who received cyclosporine, tacrolimus, mycophenolate mofetil, or thalidomide within 30 days prior to screening
14. Participants who received fecal microbial transplantation within 30 days prior to screening
15. Participants who have ever been exposed to natalizumab (Tysabri®) or oral carotegrast methyl (Carogra®)
16. Participants who received IV corticosteroids within 14 days prior to screening or during screening period
17. Participants who received therapeutic enema or suppository, other than required for colonoscopy within 14 days prior to screening or during screening
18. Screening laboratory and other analyses show abnormal results

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2027-07-21 (Estimated); Study Completion 2029-05-23 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving endoscopic response | Week 12
  Endoscopic response is defined as ≥50% reduction from baseline in centrally read Simple Endoscopic Score for Crohn's Disease (SES-CD).
  The SES-CD evaluates 4 endoscopic variables (ulcer size, ulcerated surface, affected surface, and narrowing, each on a scale from 0 (none) to 3 in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.

SECONDARY OUTCOMES:
Proportion of participants achieving clinical remission based on Crohn's Disease Activity Index (CDAI) | Week 12
  CDAI clinical remission is defined as CDAI score <150. CDAI is a composite instrument that includes participant symptoms evaluated over 7 days (abdominal pain, stool frequency and general well-being), as well as presence of complications (arthritis/arthralgia, iritis/uveitis, erythema nodosum/pyoderma gangrenosum/aphthous stomatitis, anal fissure/fistula/abscess, other fistula, and fever), the use of antidiarrheal medicines, presence of an abdominal mass, hematocrit, and body weight. These items are scored individually, weighted, and do not contribute equally to the overall score. The CDAI is derived from summing up the weighted individual scores of eight items. CDAI approximately ranges from 0 to 600 with higher scores indicating more severe disease.
Proportion of participants achieving Patient-Reported Outcome (PRO-2) remission | Week 12
  PRO 2 remission is defined as the unweighted CDAI component of daily abdominal pain (AP) score ≤1, and the unweighted CDAI component of daily average stool frequency (SF) score ≤3 (ie, AP ≤1 and SF ≤3 and no worsening from baseline).
Proportion of participants achieving both clinical remission and endoscopic response | Week 12
  Clinical remission and endoscopic response based on CDAI <150 and ≥50% reduction from baseline in centrally read Simple Endoscopic Score for Crohn's Disease (SES-CD)
Proportion of participants achieving endoscopic remission based on centrally read SES-CD | From Baseline to Week 12
  Endoscopic remission is defined as a centrally read SES-CD ≤4 points (SES-CD ≤2 points for isolated ileal disease) and a SES-CD decrease from baseline ≥2 points with no SES-CD sub score >1 point
Proportion of participants achieving CDAI clinical response | From Baseline to Week 12
  CDAI clinical response is defined as a CDAI reduction from baseline ≥100 points.
Proportion of participants achieving Inflammatory Bowel Disease Questionnaire (IBDQ) remission | Week 12
  IBDQ remission is defined as IBDQ total score ≥170 points. The Inflammatory Bowel Disease Questionnaire (IBDQ) is used to assess health-related quality of life (HRQoL) in patients with inflammatory bowel disease. It consists of 32 questions evaluating bowel and systemic symptoms, as well as emotional and social functions. Each question is answered on a scale from 1 (worst) to 7 (best). The total score ranges from 32 to 224 with higher scores indicating better health-related quality of life.
Proportion of participants achieving IBDQ response | From baseline to Week 12
  IBDQ response defined as an improvement of IBDQ scores by 27 points or more at Week 12 compared with baseline
Change from baseline in the IBDQ scores | From Baseline to week 12
  The total IBDQ score ranges from 32 to 224 which indicates better quality of life. A positive change from Baseline indicates improvement.
Plasma pre-dose concentrations of SAR441566 at selected visits | Up to week 52
Plasma post-dose concentrations of SAR441566 at selected visits | Up to week 52
Number of participants experiencing any TEAEs | Up to week 52
  Any TEAEs, including any serious opportunistic infections, psoriasiform skin lesions or other immune mediated phenomena during double-blind (DB) induction and maintenance treatment period
Number of participants experiencing any TEAEs | From week 12 to week 52
  Any TEAEs, including any serious opportunistic infections, psoriasiform skin lesions or other immune mediated phenomena during open-label treatment period

CONTACTS AND LOCATIONS:
Locations (134):
- United States (18):
  - GI Alliance - Arizona Digestive Health - Sun City- Site Number : 8400020, Sun City, Arizona
  - Bristol Hospital- Site Number : 8400007, Bristol, Connecticut
  - Novum Research- Site Number : 8400021, Clermont, Florida
  - Homestead Associates in Research- Site Number : 8400012, Homestead, Florida
  - Clinical Research of Osceola- Site Number : 8400013, Kissimmee, Florida
  - Wellness Clinical Research - Miami Lakes - 8181 Northwest 154th Street- Site Number : 8400010, Miami Lakes, Florida
  - GCP Clinical Research- Site Number : 8400004, Tampa, Florida
  - GI Alliance - Glenview- Site Number : 8400015, Glenview, Illinois
  - Illinois Gastroenterology Group- Site Number : 8400011, Gurnee, Illinois
  - University of Michigan Health System - Ann Arbor- Site Number : 8400017, Ann Arbor, Michigan
  - GI Alliance - Flowood- Site Number : 8400019, Flowood, Mississippi
  - Vector Clinical Trials- Site Number : 8400001, Las Vegas, Nevada
  - Queens Village Primary Medical Center- Site Number : 8400005, Queens Village, New York
  - Carolina Digestive Diseases and Endoscopy Center- Site Number : 8400014, Greenville, North Carolina
  - Frontier Clinical Research - Uniontown- Site Number : 8400009, Uniontown, Pennsylvania
  - Gastro Health & Nutrition- Site Number : 8400003, Katy, Texas
  - Texas Digestive Disease Consultants - Southlake- Site Number : 8400002, Southlake, Texas
  - Washington Gastroenterology - Tacoma- Site Number : 8400008, Tacoma, Washington
- Argentina (6):
  - Investigational Site Number : 0320002, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320003, Buenos Aires
  - Investigational Site Number : 0320005, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320006, Buenos Aires
- Australia (3):
  - Investigational Site Number : 0360002, Sydney, New South Wales
  - Investigational Site Number : 0360001, South Brisbane, Queensland
  - Investigational Site Number : 0360003, Parkville, Victoria
- Brazil (4):
  - Centro de Pesquisas da Clínica IBIS- Site Number : 0760001, Salvador, Estado de Bahia
  - Hospital Moinhos de Vento- Site Number : 0760006, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles- Site Number : 0760002, Porto Alegre, Rio Grande do Sul
  - Pesquisare Saude- Site Number : 0760004, Santo André, São Paulo
- Bulgaria (3):
  - Investigational Site Number : 1000001, Gorna Oryahovitsa
  - Investigational Site Number : 1000004, Sofia
  - Investigational Site Number : 1000005, Sofia
- Canada (3):
  - Investigational Site Number : 1240001, Calgary, Alberta
  - Investigational Site Number : 1240003, Montreal, Quebec
  - Investigational Site Number : 1240005, Québec, Quebec
- Chile (6):
  - Investigational Site Number : 1520007, Temuco, La Araucanía
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Viña del Mar, Región de Valparaíso
  - Investigational Site Number : 1520006, Concepción, Región del Biobío
  - Investigational Site Number : 1520004, Talcahuano, Región del Biobío
- China (12):
  - Investigational Site Number : 1560008, Changzhou
  - Investigational Site Number : 1560009, Chongqing
  - Investigational Site Number : 1560012, Fuzhou
  - Investigational Site Number : 1560001, Guangzhou
  - Investigational Site Number : 1560002, Guangzhou
  - Investigational Site Number : 1560004, Hangzhou
  - Investigational Site Number : 1560003, Hangzhou
  - Investigational Site Number : 1560007, Hefei
  - Investigational Site Number : 1560011, Nanchang
  - Investigational Site Number : 1560006, Shanghai
  - Investigational Site Number : 1560005, Shanghai
  - Investigational Site Number : 1560010, Suzhou
- Croatia (2):
  - Investigational Site Number : 1910004, Osijek
  - Investigational Site Number : 1910003, Zagreb
- Czechia (3):
  - Investigational Site Number : 2030003, Brno
  - Investigational Site Number : 2030002, Brno
  - Investigational Site Number : 2030004, Hradec Králové
- France (5):
  - Investigational Site Number : 2500005, Montpellier
  - Investigational Site Number : 2500002, Nice
  - Investigational Site Number : 2500004, Saint-Priest-en-Jarez
  - Investigational Site Number : 2500003, Toulouse
  - Investigational Site Number : 2500001, Vandœuvre-lès-Nancy
- Georgia (7):
  - Investigational Site Number : 2680006, Kutaisi
  - Investigational Site Number : 2680007, Tbilisi
  - Investigational Site Number : 2680001, Tbilisi
  - Investigational Site Number : 2680005, Tbilisi
  - Investigational Site Number : 2680002, Tbilisi
  - Investigational Site Number : 2680003, Tbilisi
  - Investigational Site Number : 2680004, Tbilisi
- Germany (5):
  - Investigational Site Number : 2760004, Berlin
  - Investigational Site Number : 2760002, Berlin
  - Investigational Site Number : 2760001, Fulda
  - Investigational Site Number : 2760005, Halle
  - Investigational Site Number : 2760006, Ludwigshafen
- Hungary (6):
  - Investigational Site Number : 3480008, Budapest
  - Investigational Site Number : 3480001, Gyöngyös
  - Investigational Site Number : 3480009, Gyöngyös
  - Investigational Site Number : 3480005, Szeged
  - Investigational Site Number : 3480006, Szekszárd
  - Investigational Site Number : 3480004, Tatabánya
- India (9):
  - Investigational Site Number : 3560007, Hyderabad
  - Investigational Site Number : 3560003, Hyderabad
  - Investigational Site Number : 3560009, Jaipur
  - Investigational Site Number : 3560001, Jaipur
  - Investigational Site Number : 3560005, Kolkata
  - Investigational Site Number : 3560006, Pune
  - Investigational Site Number : 3560002, Secunderabad
  - Investigational Site Number : 3560013, Surat
  - Investigational Site Number : 3560010, Surat
- Italy (7):
  - Investigational Site Number : 3800009, Milan, Milano
  - Investigational Site Number : 3800002, Milan, Milano
  - Investigational Site Number : 3800004, Rozzano, Milano
  - Investigational Site Number : 3800001, Padua, Padova
  - Investigational Site Number : 3800008, Rome, Roma
  - Investigational Site Number : 3800006, Rome, Roma
  - Investigational Site Number : 3800005, Pisa
- Japan (15):
  - Investigational Site Number : 3920004, Kashiwa, Chiba
  - Investigational Site Number : 3920001, Sakura, Chiba
  - Investigational Site Number : 3920005, Kitakyushu, Fukuoka
  - Investigational Site Number : 3920006, Sapporo, Hokkaido
  - Investigational Site Number : 3920010, Sapporo, Hokkaido
  - Investigational Site Number : 3920007, Sapporo, Hokkaido
  - Investigational Site Number : 3920008, Morioka, Iwate
  - Investigational Site Number : 3920019, Takamatsu, Kagawa-ken
  - Investigational Site Number : 3920020, Nagaoka, Niigata
  - Investigational Site Number : 3920003, Bunkyo, Tokyo
  - Investigational Site Number : 3920013, Hiroshima
  - Investigational Site Number : 3920002, Osaka
  - Investigational Site Number : 3920018, Ōita
  - Investigational Site Number : 3920011, Tokyo
  - Investigational Site Number : 3920012, Wakayama
- Investigational Site Number : 4800001, Vacoas, Mauritius
- Netherlands (4):
  - Investigational Site Number : 5280004, Breda
  - Investigational Site Number : 5280002, Nijmegen
  - Investigational Site Number : 5280001, Tilburg
  - Investigational Site Number : 5280003, Utrecht
- Poland (5):
  - Investigational Site Number : 6160005, Torun, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160006, Lublin, Lublin Voivodeship
  - Investigational Site Number : 6160004, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160001, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160002, Sopot, Pomeranian Voivodeship
- Romania (2):
  - Investigational Site Number : 6420004, Bucharest
  - Investigational Site Number : 6420003, Constanța
- South Korea (3):
  - Investigational Site Number : 4100002, Haeundae-Gu, Busan
  - Investigational Site Number : 4100001, Daegu, Daegu
  - Investigational Site Number : 4100003, Daejeon, Daejeon
- Spain (2):
  - Investigational Site Number : 7240002, Seville, Sevilla
  - Investigational Site Number : 7240001, Madrid
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920001, Mersin
  - Investigational Site Number : 7920002, Zonguldak

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DRI18212 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26379&tenant=MT_SNY_9011